CLINICAL TRIAL: NCT05370768
Title: Efficacy and Neurobiological Mechanisms of a Parenting-focused Mindfulness Intervention to Prevent Adolescent Substance Use
Brief Title: Parenting Mindfully Study II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Principal Investigator, Tara M. Chaplin, Ph.D., Associate Professor of Psychology, George Mason University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1770931-1
Record Dates: First submitted 2022-04-11; First posted 2022-05-12 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Adolescent Substance Use; Adolescent Psychological Symptoms; Parent Stress; Parenting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parenting Mindfully (PM) Intervention (Experimental): PM is an group based 8 week mindfulness intervention for parents.
  Interventions: Behavioral: Parenting Mindfully Intervention
- Parent Education (PE) Intervention (Active Comparator): PE is a group based 8 week educational intervention for parents that teaches parents about adolescent development.
  Interventions: Behavioral: Parenting Mindfully Intervention

INTERVENTIONS:
Behavioral: Parenting Mindfully Intervention — Includes meditation and using meditation and mindfulness in everyday life and in parenting interactions.

SUMMARY:
This study will conduct a large Randomized Controlled Trial to test effects of a parenting mindfully (PM) intervention versus a parent education (PE) intervention for highly stressed parents of adolescents.

DETAILED DESCRIPTION:
Parents of early adolescents who report experiencing stress will be randomly assigned to receive the 8 week PM or PE intervention. Before, during, and after the interventions, and at 6 month, 1 year, and 2 year follow-ups (into middle adolescence), the researchers will collect questionnaire, interview, and biological measures of parent stress, parenting, and adolescent substance use and psychological symptoms. At pre- and post-intervention, observed parenting and stress reactivity will be measured in a parent-adolescent interaction task. Some mothers will also complete fMRI sessions at pre- and post- examining emotion-related neurobiological mechanisms.

ELIGIBILITY:
Main Study Inclusion/Exclusion Criteria:

Inclusion Criteria:

1. Family with adolescent between 12-14 years;
2. High stress levels for at least one primary caregiver (referred to as "parents" throughout the application, but not required to be biological parents) on stress screener;
3. Adequate English proficiency to complete questionnaires for adolescent and at least one parent (because several of our questionnaires have not been validated for use in other languages)

Exclusion Criteria:

1. Diagnosis of intellectual disability for adolescent or psychosis for adolescent;
2. Current active suicidality that is untreated for parent or adolescent (We will refer participants with active suicidality for inpatient treatment. They will be eligible to participate in the study once stabilized),
3. Current SUDs that are untreated for parent except Tobacco Use Disorder (because participants must to be able to refrain from substances except nicotine/tobacco during the PAIT lab session day safely without withdrawal symptoms). We will refer parents with active SUDs to treatment. They will be eligible to participate in the study once stabilized and in treatment.
4. Lifetime SUD diagnosis for adolescent because an aim of the study is SUD prevention.

Note: We are recruiting for about 130 of the primary caregiver parents to be eligible in and interested in completing functional magnetic resonance imaging (fMRI) scans are pre and post-intervention. If we do not meet this number, we will restrict recruitment to those families with one parent who is interested in and eligible for fMRI.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 269 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Adolescent substance use | 2 years
  frequency and amount of substance use This will be based on combining (in a composite score) information from the Youth Risk Behavior Survey, Urine and Breath Screens, and the Timeline Follow Back Interview to determine frequency and amount of use. To combine, we will first transform all measures into z-scores (standardized scores) and then will combine them (either through composite scoring or through SEM latent variables).
Adolescent psychological symptoms | 2 years
  youth self reported symptoms on the Youth Inventory and parent reported symptoms on the Child Symptom Inventory will be combined or, if needed, tested separately in analyses. To combine, we will first transform all measures into z-scores (standardized scores) and then will combine them (either through composite scoring or through SEM latent variables).

CONTACTS AND LOCATIONS:
Locations (1):
- George Mason University, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No